CLINICAL TRIAL: NCT03423069
Title: Effects of a Diet Low in Fructose, Oligosaccharides, Disaccharides, Monosaccharides, Alcohols and Polyols in Patients With Irritable Bowel Syndrome Diarrheal Variant Respect to Dietary Advice: Randomized, Single Blind Clinical Trial.
Brief Title: Low FODMAPs Diet vs. Specific Dietary Advice in Patients With IBS Diarrheal Variant
Acronym: DIETSINIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Giuseppe Riezzo, Senior investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC2018B
Record Dates: First submitted 2018-01-22; First posted 2018-02-06 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; FODMAPs; Dietary advice; Gastrointestinal symptoms; Intestinal permeability; Gastrointestinal peptides; Microbiome; Lipidomic profile
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, single blind clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet low in FODMAPs (Experimental): Diet low in FODMAPs (diet A) during 12 weeks (with intermediate nutritional checks every 4 weeks) before returning to the final study visit.
  Interventions: Dietary Supplement: Diet low in FODMAPs
- Specific dietary advice for IBS (Active Comparator): Dietary advice for IBS (diet B) during 12 weeks (with intermediate nutritional checks every 4 weeks) before returning to the final study visit.
  Interventions: Dietary Supplement: Specific dietary advice for IBS

INTERVENTIONS:
Dietary Supplement: Diet low in FODMAPs — A strict restriction of all high FODMAP foods for the time of observation. All these foods will be identified by appropriate nutritional visits and alternatives will be suggested to ensure the diet is nutritionally adequate.
  Arms: Diet low in FODMAPs
Dietary Supplement: Specific dietary advice for IBS — Dietary recommendations such as limitation of alcohol, spicy food and fatty foods, caffeine, carbonated drinks; avoidance of chewing gums and sweeteners containing polyols; small and frequent meals; avoidance of stressful conditions and eating slowly.
  Arms: Specific dietary advice for IBS

SUMMARY:
A reduced content of FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides, and polyols) in the diet may be beneficial for patients with IBS diarrheal variant, but so far few randomized trials have reported data in favor of the effective therapeutic superiority of a low-FODMAPs diet compared to specific IBS dietary advice. On this basis, the present study is aimed, in a multidisciplinary perspective, at investigating possible changes in the symptom profile and intestinal permeability, GI peptides concentrations, metabolic and lipidomic profiles induced by these different diets in patients with IBS diarrheal variant.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional gastrointestinal disease (GI) affecting 10% -20% of the population and is composed of abdominal pain/discomfort, in combination with alterations of the stool habit. This is a functional disorder prevalent in Italy with double percentages in urban areas (13.7%) compared to rural ones (5.9%). IBS is still one of the main reasons for patients to seek for gastroenterological advice. The diagnosis of IBS is mainly based on the evaluation of symptom profiles by using different scales of assessment and also taking into account non-GI symptoms (e.g. insomnia, anxiety, and depression), as well as the characteristics of the stools. IBS is classified in different subtypes, namely: IBS diarrheal variant (IBS-D), IBS with constipation (IBS-C), IBS mixed variant (IBS-M) and non-classifiable. The pathophysiology is only partially understood and an abnormal motility, together with alterations in gut-brain communication, a low-grade inflammation, and psychosocial factors, have been variously involved. On the other hand, the therapeutic choices are still scarce. The majority of IBS subjects believe that some foods are responsible for their symptoms, tending to exclude them without, however, compromising their nutritional status [14]. Many dietary approaches have been proposed, but only a few controlled studies have been performed in this field. Recent evidence suggests that the intake of fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAPs) may trigger GI symptoms in patients with IBS. These carbohydrates are poorly absorbed in the small intestine and can pass intact in the colon, where they increase the endoluminal water through the osmotic activity and induce the production of gas due to their fermentation by intestinal bacterial flora. This, in turn, can cause abdominal distension and diarrhea. Data in the literature suggest that a diet with a reduced content in FODMAPs may be beneficial for patients with IBS and diarrhea, but so far few randomized trials have reported data in favor of the effective superiority of a low-FODMAPs diet compared to the specific dietary advice for patients with IBS. On this basis, the present study is aimed at comparing these two diets in a randomized, single-blind clinical trial in IBS patients with diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV criteria for IBS diarrhea variant (IBS-D).
* Low-lactose diet is allowed, provided that patients agree to keep this intake constant throughout the study period, except in the case of randomization in the treatment arm with a low-FODMAPs diet.
* The use of probiotic products is permitted, and patients who consume probiotic products must be instructed to continue taking the same amount previously taken throughout the study period.
* The drugs used to treat IBS, including antidepressants, will be admitted provided they are used regularly and have a stable dosage for at least one month prior to inclusion in the study.
* Patients must be willing to change their current diet to participate in the study for the whole study period.

Exclusion Criteria:

* Serious cardiac, hepatic, neurological or psychiatric diseases.
* GI diseases other than IBS (e.g., inflammatory bowel disease, celiac disease) that could explain current symptoms.
* Patients who previously had a low-content diet of particular substances (for example, low FODMAPs content, vegan diet, gluten-free diet). - This last category of subjects will be able to return to the study provided they suspend the gluten-free diet until thes symptoms reappear.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the total score of the irritable bowel syndrome - severity scoring system (IBS-SSS) questionnaire | Time frame: Before the start of the study (time 0) and after 90 days of treatment (time 90).
  IBS-SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS), leading to a total possible score of 500.
  The primary outcome corresponds to a change in the total score of the IBS-SSS questionnaire at the end of the treatment period compared to baseline, and the proportion of patients who will achieve a difference in the total symptom score of IBS-SSS ≥50 after diet. Such difference is considered a significant clinical improvement.

SECONDARY OUTCOMES:
Change in the score of the single symptom items of the irritable bowel syndrome - severity scoring system (IBS-SSS) questionnaire | Time frame: Before the start of the study (time 0) and after 90 days of treatment (time 90).
  IBS-SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS). The secondary outcome is the measure of the effects of the dietary interventions on the individual symptom items score of IBS-SSS, as well as on the characteristics of the stool habit through the administration of the diaries.
Change in the intestinal permeabily evaluation | Time frame: Before the start of the study (time 0) and after 90 days of treatment (time 90).
  For the evaluation of intestinal permeability, a test solution is prepared with 40 g sucrose (Su), 10 g lactulose (La) and 5 g mannitol (Ma) dissolved in 100 ml of water.
  The participants drink the test solution in the morning after an overnight fast and all urine samples are collected for the subsequent 5 h. Urine samples were stored at -80°C until analysis. The detection and measurement of the three sugar probes, Su, La, and Ma, in urine are performed by high-performance anion exchange chromatography coupled with pulsed amperometric detection.
Change in the GI peptide concentrations | Time frame: Before the start of the study (time 0) and after 90 days of treatment (time 90).
  To evaluate GI peptide, blood samples are collected in ice chilled tubes containing Aprotinin and EDTA. The separated plasma are stored at -70 °C until assay. Plasma levels of spexin, copeptin, meteorin, somatostatin and serotonin, are measured by enzyme immunoassay technique using commercial kits before and after the dietary interventions
Change in the lipidomic profile. | Time frame: Before the start of the study (time 0) and after 90 days of treatment (time 90).
  To evaluate the lipidomic, profile blood samples are collected in vacutainer tubes containing ethylenediaminetetraacetic acid (EDTA). The erythrocytes are separated from the plasma by centrifugation, suspended in pure water, vortexed and subsequently centrifuged to isolate the membrane pellets. Lipid extraction and lipid transesterification to fatty acid methyl esters (FAMEs) are performed using an automated protocol. Phospholipidsare will be trans-esterified to FAMEs by treatment with a potassium hydroxide (KOH)/methyl alcohol (MeOH) solution and are extracted using n-hexane. Fatty acids quantification will be performed by using a gas chromatography equipment. Quantification of fatty acid methyl esters is performed using a mixture of standards. The amount of each fatty acid is calculated before and after the dietary interventions, as a percentage of the total fatty acid content (relative %).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Russo, Principal Investigator — National Institute for Digestive Diseases IRCCS " Saverio de Bellis"
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Mearin Manrique F. Irritable bowel syndrome (IBS) subtypes: Nothing resembles less an IBS than another IBS. Rev Esp Enferm Dig. 2016 Feb;108(2):57-8. doi: 10.17235/reed.2016.4195/2016. PMID 26838485
- [Background] Gonzalez-Castro AM, Martinez C, Salvo-Romero E, Fortea M, Pardo-Camacho C, Perez-Berezo T, Alonso-Cotoner C, Santos J, Vicario M. Mucosal pathobiology and molecular signature of epithelial barrier dysfunction in the small intestine in irritable bowel syndrome. J Gastroenterol Hepatol. 2017 Jan;32(1):53-63. doi: 10.1111/jgh.13417. PMID 27087165
- [Background] Mazzawi T, El-Salhy M. Changes in duodenal enteroendocrine cells in patients with irritable bowel syndrome following dietary guidance. Exp Biol Med (Maywood). 2017 Jul;242(13):1355-1362. doi: 10.1177/1535370217699537. Epub 2017 Mar 17. PMID 28737477
- [Background] Shepherd SJ, Lomer MC, Gibson PR. Short-chain carbohydrates and functional gastrointestinal disorders. Am J Gastroenterol. 2013 May;108(5):707-17. doi: 10.1038/ajg.2013.96. Epub 2013 Apr 16. PMID 23588241
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Background] McKee AM, Prior A, Whorwell PJ. Exclusion diets in irritable bowel syndrome: are they worthwhile? J Clin Gastroenterol. 1987 Oct;9(5):526-8. doi: 10.1097/00004836-198710000-00007. PMID 3680901
- [Derived] Linsalata M, Prospero L, Ignazzi A, Riezzo G, D'Attoma B, Mallardi D, Goscilo F, Notarnicola M, De Nunzio V, Pinto G, Russo F. Depression in Diarrhea-Predominant IBS Patients: Exploring the Link Between Gut Barrier Dysfunction and Erythrocyte Polyunsaturated Fatty Acid Levels. J Clin Med. 2025 Apr 5;14(7):2483. doi: 10.3390/jcm14072483. PMID 40217932
- [Derived] Prospero L, Riezzo G, Linsalata M, Orlando A, D'Attoma B, Di Masi M, Martulli M, Russo F. Somatization in patients with predominant diarrhoea irritable bowel syndrome: the role of the intestinal barrier function and integrity. BMC Gastroenterol. 2021 May 22;21(1):235. doi: 10.1186/s12876-021-01820-7. PMID 34022802